CLINICAL TRIAL: NCT04290897
Title: A Phase II Single Arm Trial Evaluating the Safety and Efficacy of Anhydrous Enol-Oxaloacetate on Improving Cognitive Complaints in Breast Cancer Survivors
Brief Title: Oxaloacetate for the Improvement of Cognitive Complaints in Stage 0-IIIA Breast Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other); MetVital, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-001881; NCI-2020-00676 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-001881 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2020-02-25; First posted 2020-03-02 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Early-Stage Breast Carcinoma; Prognostic Stage 0 Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (anhydrous enol-oxaloacetate) (Experimental): Patients receive anhydrous enol-oxaloacetate PO BID for 8 weeks in the absence of worsening symptoms or unacceptable toxicity.
  Interventions: Drug: Anhydrous Enol-oxaloacetate; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Anhydrous Enol-oxaloacetate — Given PO
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well oxaloacetate works in reducing cognitive complaints in stage 0-IIIA breast cancer survivors. Oxaloacetate is a natural substance found in the body and is available as a nutritional supplement. Giving oxaloacetate may reduce inflammation in the brain that could be contributing to cognitive complaints seen after cancer treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the effectiveness of anhydrous enol-oxaloacetate (oxaloacetate) in reducing cognitive complaints in breast cancer patients over the course of 8 weeks.

SECONDARY OBJECTIVES:

I. To assess the tolerability of oxaloacetate. II. To examine whether oxaloacetate has an effect on the neurocognitive domain of executive function.

III. To examine whether oxaloacetate has an effect on patient reported fatigue, insomnia, and depressive symptoms.

IV. To collect blood for assessment of inflammatory markers and glutamate levels.

OUTLINE:

Patients receive anhydrous enol-oxaloacetate orally (PO) twice daily (BID) for 8 weeks in the absence of worsening symptoms or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women with a diagnosis of early stage breast cancer (stage 0, I, II, IIIa) who are at least 12 months after surgery, chemotherapy, radiation, but may be on endocrine therapy or HER-2 targeted therapy, and not more than 5 years after their breast cancer diagnosis
* No evidence of active/recurrent breast cancer or other serious chronic illness
* Has significant cognitive complaints, defined as a score of < 12 on the Patient-Reported Outcomes Measurement Information System (PROMIS) Adult version (v) 2.0 - Cognitive Function 4a
* Is geographically accessible, and able to participate in a study of 8-10 weeks duration
* Ability to complete evaluation surveys in English
* The effects of oxaloacetate on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of childbearing potential must agree to use adequate contraception (barrier method of birth control; intrauterine device [IUD]; abstinence) prior to study entry and for the duration of study participation. Women of any age who have had their ovaries and/or uterus removed will not be at risk for pregnancy and will not require contraception. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately. Menopausal status will be established as follows: Women who are 55 years or older and who are not menstruating will be considered postmenopausal and not at risk for pregnancy. Women who are less than 55 years old who are menstruating will be considered premenopausal and will require contraception. Women who are less than 55 years with an intact uterus and ovaries who are not menstruating and have not had a menstrual period within the past 2 years will have an follicle-stimulating hormone (FSH) and estradiol measured. If the values are in postmenopausal range the woman will be considered postmenopausal and she will not be considered at risk for pregnancy
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Has another serious or chronic medical or psychiatric condition that contributes to substantial physical or emotional disability that would detract from participating in the planned study
* Taking chronic medications that would interfere with cognitive functioning such as medications for sleep, anxiety, narcotics for pain, use of illicit drugs or cannabis
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to oxaloacetate
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast-feeding women are excluded from this study because the safety of oxaloacetate in this setting is unknown. A pregnancy test will be performed on all women with an intact uterus and ovaries who are not determined to be postmenopausal

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy-Cognitive Function Perceived Cognitive Impairment (FACT-Cog PCI) score | Baseline up to day 57
  Patients who have an improvement in the FACT-Cog PCI of at least 4 points will be considered to have a positive response. The response proportion will be further characterized using a point estimate and 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to day 57
  Will be assessed by Common Terminology Criteria for Adverse Events version 4.
Fatigue | At day 57
  Will be assessed by Multidimensional Fatigue Symptom Inventory. Scores will be summarized as means and standard deviations and confidence intervals will be calculated. Changes will also be summarized as effect sizes to support design of a future trial.
Insomnia | At day 57
  Will be assessed by the Insomnia Severity Index. Scores will be summarized as means and standard deviations and confidence intervals will be calculated. Changes will also be summarized as effect sizes to support design of a future trial.
Depressive symptoms | At day 57
  Will be assessed by Patient-Reported Outcomes Measurement Information System. Scores will be summarized as means and standard deviations and confidence intervals will be calculated. Changes will also be summarized as effect sizes to support design of a future trial.
Neurocognitive tests | Up to day 57
  Subjects will be assessed by the California Verbal Learning Test-2nd edition, Brief Visuospatial Memory Test-Revised, Golden Stroop, Trail Making Test, Verbal Fluency, Connor's Continuous Performance Test-II. All scales listed will have the individual scores transformed by using published normative data, therefore the unit of measure will be the same for the listed tests; higher scores indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Ganz, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States